CLINICAL TRIAL: NCT02634814
Title: Improving Disability in Knee Osteoarthritis by Targeting Neuromuscular Deficits
Brief Title: The KNEEhabilitation Study: Improving Disability in Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-1150
Record Dates: First submitted 2015-12-03; First posted 2015-12-18 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Transcutaneous Electric Nerve Stimulation; Exercise Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TENS and Therapeutic Exercise (Experimental): Patients assigned to the TENS+Therapeutic Exercise (TE) group will receive a Select System TENS unit (EMPI, Inc., St. Paul, MN), and 8 hours of TENS per day (150 pulses per second, 150 msec phase duration at a patient-perceived strong sensory intensity). Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist. Each TE Session will last 45 minutes and include open and closed chain lower extremity muscle strengthening exercises. The exercise will be progressed using the Daily Adjusted Progressive Resistive Exercise Program.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Other: Therapeutic Exercise
- Sham TENS and Therapeutic Exercise (Sham Comparator): Sham TENS+TE patients will receive a Select System TENS unit (EMPI, Inc., St. Paul, MN) specifically configured to cease TENS current output 20 seconds after the participants initiation. For blinding purposes, patients will be told that they should feel a brief stimulation (~20 seconds) that will become "sub-sensory" in nature. The participants will wear the Sham TENS for 8 hours per day. Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist. Each TE Session will last 45 minutes and include open and closed chain lower extremity muscle strengthening exercises. The exercise will be progressed using the Daily Adjusted Progressive Resistive Exercise Program.
  Interventions: Other: Therapeutic Exercise; Device: Sham Transcutaneous Electrical Nerve Stimulation
- Therapeutic Exercise Only (Active Comparator): The role of the comparison group is to provide data on how traditional TE affects the outcome measures. The TE only group will allow us to assess how the addition of TENS to traditional TE will augment the effects of traditional TE. Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist. Each TE Session will last 45 minutes and include open and closed chain lower extremity muscle strengthening exercises. The exercise will be progressed using the Daily Adjusted Progressive Resistive Exercise Program.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — TENS is FDA approved for the purposes in which we will be applying the modality (21CFR882.5890; http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/cfrsearch.cfm?fr=882.5890, these TENS Units have been acquired by the PI, who is a licensed Allied Health Professional in the state of North Carolina).
  Other Names: TENS
  Arms: TENS and Therapeutic Exercise
Other: Therapeutic Exercise — Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist. Each TE Session will last 45 minutes and include open and closed chain lower extremity muscle strengthening exercises. The exercise will be progressed using the Daily Adjusted Progressive Resistive Exercise Program. The intervention will consist of 10 45-minute sessions.
  Other Names: Physical Therapy
Device: Sham Transcutaneous Electrical Nerve Stimulation — Sham TENS+TE patients will receive a Select System TENS unit (EMPI, Inc., St. Paul, MN) specifically configured to cease TENS current output 20 seconds after the participants initiation. For blinding purposes, patients will be told that they should feel a brief stimulation (~20 seconds) that will become "sub-sensory" in nature. The participants will wear the Sham TENS for 8 hours per day.
  Arms: Sham TENS and Therapeutic Exercise

SUMMARY:
The focus of this project is to use transcutaneous electrical nerve stimulation (TENS) for the novel indication of treating neuromuscular activation in individuals with knee osteoarthritis (OA) that exhibit neuromuscular activation deficits. The overall goal is to improve outcomes associated traditional therapeutic exercise (TE) by developing an enhanced rehabilitation strategy, which augments TE with TENS (TENS+TE), for the purpose of treating underlying neuromuscular activation deficits. The investigators seek to use TENS to excite neural pathways that immediately increase neuromuscular activation as well as cause sustained improvements in neuromuscular activation and greater strength gains in knee OA patients compared to traditional TE. The investigators will evaluate the effect of TENS+TE on muscle strength, neuromuscular activation, gait biomechanics, physical function, physical activity, self-efficacy of physical activity, self-reported quality of life, disability and pain. The central hypothesis is that an enhanced TENS+TE intervention will lead to better clinical outcomes, increased physical activity, and improved general health. The rationale for conducting a small clinical trial, which demonstrates the feasibility and establishes the preliminary effects of an enhanced rehabilitation strategy, is ultimately to inform the development of a future larger clinical trial to establish the efficacy of an enhanced rehabilitation strategy for knee OA. This hypothesis will be tested through two specific aims: 1) to collect and report data on the feasibility of conducting a clinical trial to evaluate the efficacy of using TENS+TE compared to sham TENS+TE and to TE only for treating patients with knee OA in a clinical setting, and 2) to determine preliminary effects of a 4-week TENS+TE intervention compared to sham TENS+TE, and TE only on muscle strength, neuromuscular activation, gait biomechanics, physical function, physical activity, self-efficacy of physical activity, self reported quality of life, disability, and pain in knee OA patients. Posttests will be at 4 and 8-weeks following baseline.

ELIGIBILITY:
Inclusion Criteria:

* All knee OA participants must exhibit symptomatic knee OA, which we will define as a normalized, person based, Western Ontario and McMaster Universities Arthritis Index (WOMAC) function subscale score > 31 (out of 100 points, indicating most dysfunction),38 radiographic evidence of tibiofemoral OA (2-4 on the Kellgren - Lawrence scale) 39 and neuromuscular activation deficits, defined as quadriceps neuromuscular activation of less than 90% in the involved leg.3 Participants between the ages of 40 and 75 years old will be included.

Exclusion Criteria:

* Patients will also be excluded if they have: 1) been diagnosed with a cardiovascular condition restricting exercise; 2) had a corticosteroid or hyaluronic acid injection in the involved knee in the previous 6-months; 3) a pacemaker; 4) a neurodegenerative condition; 5) rheumatoid arthritis; 6) cancer; 7) neural sensory dysfunction over the knee 8) a BMI over 35; 9) history of lower extremity orthopaedic surgery in the past year; 10) a history of a traumatic knee injury in the past 6 months; 11) any history of a total knee arthroplasty in either extremity; or 12) a diagnosed, non-reconstructed knee ligament tear. Patients needing an assistive device to walk and pregnant females will also be excluded.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pietrosimone, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TENS and Therapeutic Exercise: Patients assigned to this group will receive a Select System TENS (i.e., transcutaneous electrical nerve stimulation TENS) unit, and 8 hours of TENS per day (150 pulses per second, 150 msec phase duration at a patient-perceived strong sensory intensity). Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist.
- Sham TENS and Therapeutic Exercise: Patients will receive a Select System TENS unit specifically configured to cease TENS current output 20 seconds after the participants initiation. For blinding purposes, patients will be told that they should feel a brief stimulation (~20 seconds) that will become "sub-sensory" in nature. The participants will wear the Sham TENS for 8 hours per day. Ten sessions of traditional therapeutic exercise (TE) will be provided under the supervision of a licensed Physical Therapist. Each TE Session will last 45 minutes and include open and closed chain lower extremity muscle strengthening exercises. The exercise will be progressed using the Daily Adjusted Progressive Resistive Exercise Program.
- Therapeutic Exercise Only: Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist. Each TE Session will last 45 minutes and include open and closed chain lower extremity muscle strengthening exercises. The exercise will be progressed using the Daily Adjusted Progressive Resistive Exercise Program.
Period: Overall Study
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only
Started | 32 | 29 | 29
Completed | 30 | 23 | 29
Not Completed | 2 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- TENS and Therapeutic Exercise: Patients assigned to this group will receive a Select System TENS unit, and 8 hours of TENS per day (150 pulses per second, 150 msec phase duration at a patient-perceived strong sensory intensity). Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist.
- Sham TENS and Therapeutic Exercise: Patients will receive a Select System TENS unit specifically configured to cease TENS current output 20 seconds after the participants initiation. For blinding purposes, patients will be told that they should feel a brief stimulation (~20 seconds) that will become "sub-sensory" in nature. The participants will wear the Sham TENS for 8 hours per day. Ten sessions of TE will be provided under the supervision of a licensed Physical Therapist. Each TE Session will last 45 minutes and include open and closed chain lower extremity muscle strengthening exercises. The exercise will be progressed using the Daily Adjusted Progressive Resistive Exercise Program.
- Total: Total of all reporting groups
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only | Total
Number analyzed (Participants) | 32 | 29 | 29 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 21 | 22 | 68
  >=65 years | 7 | 8 | 7 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 14 | 51
  Male | 14 | 10 | 15 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 6 | 19
  White | 25 | 23 | 22 | 70
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 29 | 29 | 90

OUTCOME MEASURES:

1. Primary Outcome: Mean in Self-reported Disability Score as Measured by the Western Ontario and McMasters Universities Index Between Groups
Description: The Western Ontario and McMasters Universities Index is reliable and valid measure of self reported disability. The physical function consists of 17 items and asks about the magnitude of difficulty when ascending and descending stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on and taking off socks, rising from bed, lying in bed, getting in and out of the bath, sitting, getting on and off the toilet, completing heavy household duties, and completing light household duties. Each item is presented in a 5 point Likert-type format and uses the following descriptors for possible answer choices none, mild moderate, severe, and extreme. Each descriptor corresponds to an ordinal scale of 0-4. The scores are summed for the items in each subscale, with total possible ranges as 0-68. Higher scores on the WOMAC indicate greater amounts of functional limitations.
Time Frame: 8-weeks from Baseline
Population: A proportion of the participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only
Number analyzed (Participants) | 30 | 23 | 29
score on a scale | 20.6 (11.91) | 20.57 (11.54) | 21.72 (9.80)

2. Primary Outcome: Mean Voluntary Quadriceps Activation as Measured by the Central Activation Ratio Expressed as a Percent of Full Activation
Description: The investigators assessed voluntary quadriceps central activation ratio as a representative variable of lower extremity neuromuscular activation using the supra imposition technique. Quadriceps central activation ratio has been demonstrated to be significantly decreased in knee osteoarthritis (OA) compared to healthy, matched controls, and the investigators have reported acceptable measurement reliability (ICC2,k = 0.85)
Time Frame: 8-weeks from Baseline
Population: Difference in baseline individuals and number of participants are due to a proportion of patients lost to follow up and participants electing not to undergo voluntary quadriceps activation.
Measure: Mean (Standard Deviation); unit: percentage of full activation
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only
Number analyzed (Participants) | 26 | 27 | 27
percentage of full activation | 87.5 (9.9) | 85.8 (12.5) | 86.7 (11.8)

3. Primary Outcome: Mean Maximal Quadriceps Strength as Measured by the Maximal Isometric Voluntary Contractions Normalized to Body Weight
Description: Quadriceps strength was measured in Newton Meters normalized to body weight of the individuals. Strength was assessed in 90 degrees of knee flexion.
Time Frame: 8-weeks from Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nm/kg body weight
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only
Number analyzed (Participants) | 29 | 22 | 27
Nm/kg body weight | 1.5 (0.58) | 1.53 (0.48) | 1.54 (0.57)

4. Primary Outcome: Mean Internal Knee Extension Moment During Walking Gait Measured in Nm/ Body Weight*m
Description: The peak internal knee extension moment was calculated using using inverse dynamics calculations in the first 50% of the stance phase of gait and normalized to the Body Weight* height (m) of the individual during self selected gait speed.
Time Frame: 8-weeks from Baseline
Population: Difference in baseline individuals and number of participants are due to a proportion of patients lost to follow up and measurable outcomes were unable to be analyzed due to error in positioning of knee joint center marker.
Measure: Mean (Standard Deviation); unit: Nm/ Body Weight *m
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only
Number analyzed (Participants) | 18 | 16 | 23
Nm/ Body Weight *m | .027 (.015) | .03 (.015) | .029 (.013)

5. Primary Outcome: Mean Knee Flexion Angle During Walking Gait Measured in Degrees of Knee Flexion
Description: The peak Knee Flexion Angle was calculated using using inverse dynamics calculations in the first 50% of the stance phase of gait and during self selected gait speed.
Time Frame: 8-weeks from Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only
Number analyzed (Participants) | 18 | 16 | 23
degrees | 9.97 (7.39) | 9.05 (5.75) | 9.3 (5.75)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through 8 weeks following Baseline.
Arm/Group | TENS and Therapeutic Exercise | Sham TENS and Therapeutic Exercise | Therapeutic Exercise Only
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/32 | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02634814/Prot_SAP_000.pdf